CLINICAL TRIAL: NCT05457894
Title: Randomized, Double-blind, Comparative, Controlled Trial of Tolerability, Reactogenicity, Safety and Immunogenicity of Flu-M [Inactivated Split Influenza Vaccine] in Pregnant Women During the 2nd - 3rd Trimester
Brief Title: Trial of Tolerability, Reactogenicity, Safety and Immunogenicity of Flu-M [Inactivated Split Influenza Vaccine] in Pregnant Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St. Petersburg Research Institute of Vaccines and Sera (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FM-2019-01
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Influenza, Human; Vaccination; Infection; Vaccines
Keywords: Influenza; Flu; Vaccine; FLU-M; SPbSRIVS; Ultrix
MeSH Terms: conditions — Influenza, Human; Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Flu-M, II trimester of pregnancy (Experimental): Subjects during their II trimester of pregnancy (gestational age: 14-26 weeks), immunized once with the Flu-M vaccine.
  Interventions: Biological: Flu-M, Inactivated split influenza vaccine
- Ultrix®, II trimester of pregnancy (Active Comparator): Subjects during their II trimester of pregnancy (gestational age: 14-26 weeks), immunized once with Ultrix®.
  Interventions: Biological: Ultrix®, Inactivated Split Influenza Vaccine
- Flu-M, III trimester of pregnancy (Experimental): Subjects during their III trimester of pregnancy (gestational age: 27-32 weeks), will be immunized once with the Flu-M vaccine.
  Interventions: Biological: Flu-M, Inactivated split influenza vaccine
- Ultrix®, III trimester of pregnancy (Active Comparator): Subjects during their III trimester of pregnancy (gestational age: 27-32 weeks), immunized once with Ultrix®.
  Interventions: Biological: Ultrix®, Inactivated Split Influenza Vaccine

INTERVENTIONS:
Biological: Flu-M, Inactivated split influenza vaccine — solution for intramuscular injection, 0.5 ml
  Arms: Flu-M, II trimester of pregnancy; Flu-M, III trimester of pregnancy
Biological: Ultrix®, Inactivated Split Influenza Vaccine — solution for intramuscular injection, 0.5 ml
  Arms: Ultrix®, II trimester of pregnancy; Ultrix®, III trimester of pregnancy

SUMMARY:
Comparative study of tolerability, reactogenicity, safety and immunogenicity Flu-M [Inactivated Split Influenza Vaccine] vs. the Ultrix® vaccine for the prevention of influenza in pregnant women in the 2nd-3rd trimesters of pregnancy

DETAILED DESCRIPTION:
This is a randomized, double-blind, comparative, controlled trial. A design with a control group treated with Ultrix®, inactivated influenza vaccine, was chosen to obtain objective findings.Trial population: healthy women aged 18 to 35 years during the 2nd and 3rd trimesters of pregnancy. Subjects were randomized into 4 groups in a ratio of 1:1:1:1, 50 subjects per group.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of signed Informed Consent of the female patient to participate in the trial
2. Healthy women aged 18 to 35 years in their 2nd and 3rd trimesters of pregnancy with gestational age of no more than 32 weeks
3. Singleton pregnancy progressing normally
4. No contraindications for vaccination
5. Pregnant women that are able to fulfill the requirements of the protocol (i.e., fill out the Self-Observation Diary, come to follow-up visits)
6. The investigator is given the opportunity to collect data about somatic, infectious, and allergic diseases within at least 3 months from vaccination (one or more calls from the clinical investigator or visits per month (as needed))

Exclusion Criteria:

1. Body temperature above 37°С
2. History of influenza or previous influenza vaccination during 6 months before the screening
3. History of allergic reactions to chicken protein
4. Allergic reactions to vaccine components or any previous vaccination
5. Gestational toxicosis
6. Any disorders of pregnancy
7. Thyroid disorders
8. Bronchial asthma
9. Clotting disorders
10. 1, 2 type diabetes mellitus
11. High risk of fetal chromosomal abnormalities (individual risk of at least 1/100) in the 1st trimester of pregnancy and/or the detection of fetal congenital anomalies / developmental defects in the 1st, 2nd, and 3rd trimesters of pregnancy
12. Strong reaction (temperature above 40 °C, hyperemia or edema more than 8 cm in diameter) or complications (collapse or shock-like condition) that developed within 48 hours from prior vaccination; convulsions accompanied or not accompanied by a fever due to any prior vaccination
13. Acute infectious or non-infectious diseases less than 4 weeks before the screening, exacerbation of chronic diseases (the vaccination can be carried out after recovery or in the period of remission)
14. Immunomodulatory therapy, including immune-enhancing, immunosuppressive therapy (corticosteroids, cytotoxic and radioactive drugs) in the 6 months preceding the trial
15. Any other contraindications against vaccination according to the investigator.
16. Leukemia, cancer or a positive reaction to HIV infection, hepatitis B and C, syphilis in the medical history
17. Volunteers who received immunoglobulin or blood products within the last three months before the trial
18. History of Guillain-Barré syndrome (acute polyneuropathy)
19. Autoimmune diseases
20. Any confirmed or suspected immunosuppressive or immunodeficiency condition
21. Respiratory, cardiovascular failure, impaired liver or kidney function.
22. Severe birth defects or serious chronic diseases, including any clinically significant chronic diseases of lungs, kidneys, cardiovascular, nervous system, psychiatric diseases or metabolic disorders, confirmed by medical history or objective examination
23. Vaccination with any vaccine less than 30 days before the screening or scheduled vaccination with any vaccine within 30 days from vaccination with the trial vaccines
24. The woman is/was a patient of a tuberculosis dispensary and/or narcological dispensary and/or neuropsychiatric dispensary
25. Chronic alcohol abuse and/or use of drugs in the past history
26. Smoking
27. Participation in another clinical trial during the last 3 months

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Healthy women aged 18 to 35 years during the 2nd and 3rd trimesters of pregnancy.
Enrollment: 207 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Seroprotection rate at day 21 after vaccination | Days 0 (screening), 21
  The percentage of vaccinees who have an antibody titer of more than 1:40 by Day 21 after vaccination.
  Antibodies to influenza B, А (H1N1), А (H3N2) viruses Seroprotection rate ≥ 70%.
Change from Baseline Seroconversion rate at day 21 after vaccination | Days 0 (screening), 21
  The relative number of vaccinees, whose titer of hemagglutinin inhibiting antibodies has increased by more than 4 times vs. baseline among all immunoprotective persons.
  Antibodies to influenza B, А (H1N1), А (H3N2) viruses Seroconversion rate ≥ 40%
Change from Baseline Seroconversion factor at day 21 after vaccination | Days 0 (screening), 21
  An increase in the geometric mean titers of hemagglutinin inhibiting antibodies on Day 21 vs. baseline, expressed in multiplicity of increase.
  Antibodies to influenza B, А (H1N1), А (H3N2) viruses Seroconversion factor ≥ 2.5

SECONDARY OUTCOMES:
Incidence of AEs and SAEs associated with vaccination | Day 1 (30 minutes, 3 and 5 hours after vaccination), days 2-21
  The degree of intensity or severity of AE was evaluated on a 4-point scale:
  0 - none (no symptoms)
  1. - mild (mild symptoms)
  2. - moderate (symptoms that disrupt normal daily activities to a certain extent)
  3. - severe (symptoms that disrupt normal daily activities)
Number of participants with abnormal changes in physical examination data | Days 0-7, day 21
  Physical examination includes examination of the general appearance, condition of the skin and mucous membranes, neck (including the thyroid gland), eyes, ears, nasopharynx, lungs, heart, abdomen, liver, back, lymph nodes Table 6
Number of participants with abnormal changes in vital signs - Blood pressure (BP) | Days 0-7, day 21
  BP is measured in a sitting position after 10 minutes of rest
Number of participants with abnormal changes in vital signs - Heart rate (HR) | Days 0-7, day 21
  HR is measured in a sitting position after 10 minutes of rest
Number of participants with abnormal changes in vital signs - Respiratory rate (RR) | Days 0-7, day 21
  RR is measured in a sitting position after 10 minutes of rest
Number of participants with abnormal changes in vital signs - Body temperature | Days 0, 1 (10 minutes before vaccination, 30 minutes and 2 and 5 hours after vaccination), days 2-7, day 21
  Body temperature is measured in the armpit
Incidence and severity of systemic post-injection reactions | Day 1 (30 minutes, 3 and 5 hours after vaccination), days 2-21
Incidence and severity of local post-injection reactions | Day 1 (30 minutes, 3 and 5 hours after vaccination), days 2-21
Number of participants with abnormal changes data obtained from examinations by immunologist-allergist | Days 1-7, day 21
  Number of participants with clinically significant abnormalities
Number of participants with abnormal changes of neurological examination data | Days 0-7, day 21
  Number of participants with clinically significant abnormalities
Number of participants with abnormal changes data obtained from examinations by obstetrician-gynecologist | Days 0-7, day 21
  Examination: Respiratory organs, Blood circulation organs, Digestive organs, Organs of the urinary system, Mammary glands, Tone of the uterus, Fetal palpation results, Fetal auscultation results
Number of participants with abnormal changes in the ultrasound data assessment of fetus and uterus | Days 0 (screening), 21
Number of participants with clinically significant abnormalities - Complete blood count (CBC) | Days 0 (screening), 3, 21
  Red cells, Hemoglobin, ESR, White cells, Platelets, Relating to stab neutrophile, Segmented neutrophils, Lymphocytes, Eosinophils, Basophils, Monocytes
Number of participants with clinically significant abnormalities - Biochemical blood test (BBT) | Days 0 (screening), 3, 21
  Creatinine, Urea, Aspartate aminotransferase (AST), Alanine transaminase (ALT), Lactate dehydrogenase (LDH), Total protein, C-reactive protein, Alkaline phosphatase, Bilirubin, Glucose, Cholesterol, Prothrombin complex, Thymol test, β-lipoproteins
Number of participants with clinically significant abnormalities - Urinalysis | Days 0 (screening), 3, 21
  Density, Leukocytes, pH, color, urine glucose, urine erythrocytes, bacteria
Number of participants with abnormal changes of total IgE | Days 0 (screening), 3, 21

CONTACTS AND LOCATIONS:
Overall Officials: Ellina Ruzanova, PhD, Study Director — St. Petersburg Research Institute of Vaccines and Sera
Locations (5):
- Russia (5):
  - Federal State Budgetary Educational Institution of Higher Education "Altai State Medical University" of the Ministry of Health of the Russian Federation, Barnaul, Altai Territory
  - Federal State Budgetary Institution "Siberian Federal Scientific and Clinical Center of Federal Medical and Biologic Agency", Seversk, Tomsk Oblast
  - "Curator" Limited Liability Company, Saint Petersburg
  - KOROLEV MEDICINE Limited Liability Company, Saint Petersburg
  - Municipal Budgetary Institution "Central City Hospital No.7", Yekaterinburg